CLINICAL TRIAL: NCT01247506
Title: Identification of Survival-related microRNAs in Hepatocellular Carcinoma
Brief Title: Different Genetic Features Associated With Hepatic Carcinogenesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Po-Huang Lee, Proferrsor, Department of sugery, National Taiwan University Hospital
Other Study IDs: 200912020R
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: microRNA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — HCC tissues and paired nontumor tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: tumor tissues of HCC patients
- 2: paired nontumor tissues of HCC patients

SUMMARY:
The purpose of this study is to identify different genetic features in hepatocellular carcinoma. It will assist in predicting individual risks of disease progression and would help to clarify pathophysiological mechanisms of HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a leading cause of cancer deaths in Taiwan. HCC normally develops as a consequence of underlying liver disease and is most often associated with cirrhosis. Surgical resection and liver transplantation are current best curative options to treat HCC. However, recurrence or metastasis is quite common in patients who have had a resection and survival rate is 30% to 40% at 5 years postoperatively.

MicroRNAs, small non-coding RNA, act as endogenous RNA interference by post-transcription regulation. Recent studies suggest that microRNAs may act as tumor suppressors or oncogenes and altered microRNA expression levels may play an important role in the cancer initiation and progression. Several studies, including ourselves, have shown that specific microRNAs are aberrantly expressed in malignant HCC tissues compared to normal counterpart. Although many microRNA profiling studies were done to diagnose hepatocarcinogenesis, data about prognostic significances for postsurgical survival are very limited. The main point of this study is to develop a predictive signature for postsurgical survival in HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hepatocellular carcinoma

Exclusion Criteria:

-

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 160 patients with histologically proven HCC were collected by Dr. Po-Huang Lee's Lab (The Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Po-Huang Lee, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan